CLINICAL TRIAL: NCT04446884
Title: Treatment of Stress Urinary Incontinence in Women With Autologous Adipose-derived Mesenchymal Stem Cells Mixed With Collagen Gel
Brief Title: Treatment of Stress Urinary Incontinence in Women With Autologous Adipose-derived Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_MSC(UIW)
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; Mesenchymal stem cells
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cells (Experimental): Patients with Stress urinary incontinence receiving standard treatment plus adipose-derived mesenchymal stem cells
  Interventions: Biological: Autologous adipose-derived mesenchymal stem cells; Other: Standard treatment according to the Clinical protocols
- control (Active Comparator): Patients with Stress urinary incontinence receiving standard treatment
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: Autologous adipose-derived mesenchymal stem cells — Autologous adipose-derived mesenchymal stem cells mixed with collagen solution
  Arms: mesenchymal stem cells
Other: Standard treatment according to the Clinical protocols — Standard treatment according to the Clinical protocols

SUMMARY:
Treatment of women with stress urinary incontinence using injection of autologous adipose-derived mesenchymal stem cells mixed with collagen gel

DETAILED DESCRIPTION:
During the implementation of the project, method for the treatment of women stress urinary incontinence using injection of autologous adipose-derived mesenchymal stem cells mixed with collagen was developed.

Effectiveness of MSCs is due to the following:

* the ability of MSCs to stimulate tissue regeneration
* positive results of preclinical studies of the method of treatment of stress urinary incontinence (SUI) in animals (female rats).

After gynecological examination, diagnosis of SUI, MSCs were isolated from adipose tissue, cultured and then transplanted back to directly under mucosa of urethra by three point injection in one third distal from the urethral neck at 3, 6 and 9 o'clock and to the paraurethral area.

Injected volume was 3 ml per patient. For injection MSCs (6*10^6 cells) were mixed with collagen solution (3,5% w|w).

Follow up patients monitoring was mperformed at 2, 4, 6 and 12 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Stress urinary incontinence
* absence of acute inflammatory manifestations in the genitourinary system

Exclusion Criteria:

* urethral or bladder malformations
* acute and chronic infectious diseases: HIV, viral hepatitis, tuberculosis
* mental disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of cured patients | 3 months
  Number of patients cured
Number of patients with treatment-related adverse events | 4 weeks
  MSC application related adverse events assessed by blood count, liver and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor D Volotovski, Prof, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Alexander Nechiporenko, Dr, Study Director — Associate Professor of Department of Surgical Diseases
Locations (1):
- Hrodna City Clinical Hospital, Hrodna, Belarus

IPD SHARING:
Plan to Share IPD: No